CLINICAL TRIAL: NCT03447067
Title: Computer Guided Versus Conventional Surgical Removal of Deeply Impacted Mandibular Third Molar With Preservation of External Oblique Ridge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alaadden Mahmoud Abu Al Enein (Other)
Responsible Party: Sponsor-Investigator, Alaadden Mahmoud Abu Al Enein, Principal Investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 171986
Record Dates: First submitted 2018-02-10; First posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Impacted Third Molar Tooth

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional surgery (Experimental): comprised 9 patient undergoing surgical removal of deeply impacted mandibular third molar by regular manor.
  (Based on :Panorama and CBCT ) technique : 1- flap design 2- bone removal 3- tooth division 4- closure flap (suture)
  Interventions: Procedure: computer guided surgical; Device: CBCT
- computer guided surgery (Experimental): comprised 9 patient undergoing surgical removal of deeply impacted mandibular third molar using computer guided surgical cutting stent.
  Based on (panorama , CBCT and fabricating computer guided stent technique: 1- flap design 2- accurate setting stent in a predesign site 3- bony window removing according to the stent design 4- surgical separation of the teeth with extraction the remaning part . 5- identify the nerve 6- replace the bony window in to original place with stability 7- closure and depridment
  Interventions: Procedure: Conventional surgery; Device: CBCT

INTERVENTIONS:
Procedure: computer guided surgical — has three cutting guided plane for identify the position of place of the third molar, it have beveled cut for stability after remove the teeth and placing the bony window
  Arms: Conventional surgery
Procedure: Conventional surgery — Low speed motor with surgiacl round burs and surgical fissure for removal a covering bone with decapitation and guttering formation
  Arms: computer guided surgery
Device: CBCT — For measuring the bone removeal
  Arms: Conventional surgery
Device: CBCT — for identifed the nerve
  Arms: computer guided surgery

SUMMARY:
in patent have deeply impacted lower third molar ,dose computer guided enhance surgical outcome versus conventional surgical remove of wisdom teeth

DETAILED DESCRIPTION:
P- Patient with deeply impacted mandibular molar I- Computer guided surgical cutting stent C- Conventional extraction O- Clinical outcome sound radiographic outcomes primary outcome

- pain : each patient well be asked to rate current and worst pain intensity on visual analogue scale (VAS ) of 0-10 with Zero being no pain and Ten corresponds to the worst pain.

Secondary outcome

* evaluation of maximum inter incisal opening: assessment of MMO will be performed by measuring the distance in mm between the incisal edges of the upper and lower central incisor by using tape graduated method.
* evaluation of edema throw use nylon thread.

ELIGIBILITY:
Inclusion Criteria:

* patient with deeply impacted mandibular third molar
* patients should be free from any systematic disease that affect normal healing

Exclusion Criteria:

* -Patient with soft tissue impaction and impaction class A position 1
* Medical problem that may interfere with the procedures such as bleeding disorder & pregnant.
* Uncooperative patient.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-03-28 (Estimated); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
Pain | immediate post operative ,at three day pain change till fourteen day day .
  each patient well be asked to rate current and worst pain intensity on visual analogue scale (VAS ) of 0-10 with Zero being no pain and Ten corresponds to the worst pain(pain change during follow up period .

SECONDARY OUTCOMES:
evaluation of maximum inter incisal opening | immediate post operative ,at three day inter incisal change till fourteen day .
  assessment of MMO will be performed by measuring the distance in mm between the incisal edges of the upper and lower central incisor by using tape graduated method.

IPD SHARING:
Plan to Share IPD: Undecided